CLINICAL TRIAL: NCT04020094
Title: Perioperative Atezolizumab With MVA-BN-Brachyury and PROSTVAC For Intermediate-Risk And High-Risk Localized Prostate Cancer
Acronym: AtezoVax
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding source withdrawn
Sponsor: University of Utah (Other)
Collaborators: Bavarian Nordic (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI121075
Record Dates: First submitted 2019-07-08; First posted 2019-07-15 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Prostate Adenocarcinoma
Keywords: intermediate-risk prostate cancer; high-risk prostate cancer; very high-risk prostate cancer
MeSH Terms: interventions — PROSTVAC; atezolizumab

STUDY DESIGN:
Intervention Model Description: This study is a prospective, open label, single arm phase II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental)
  Interventions: Combination Product: MVA-BN-Brachyury

INTERVENTIONS:
Combination Product: MVA-BN-Brachyury — Cycle= 21 days. Neoadjuvant Therapy: Treatment will be given for 2 neoadjuvant cycles. MVA-BN-Brachyury will be administered as intratumoral injection on Day 1 of each of 2 neoadjuvant cycles. PROSTVAC-V will be administered as a subq injection on Day 1 of Cycle 1 (the first neoadjuvant cycle) and PROSTVAC-F will be administered as a subq injection on Day 1 of Cycle 2 (the second neoadjuvant cycle). Atezolizumab will be given as an infusion on Day 1 of each 2 neoadjuvant cycles.
  MVA-BN-Brachyury will be injected intratumorally into the prostate. Injections will target PI-RADS 4 and 5 lesions.
  Surgery: Patients will undergo SOC radical prostatectomy Adjuvant Therapy: Systemic treatment with atezolizumab and PROSTVAC-F will be reinitiated between 3 to 8 weeks after surgery and will continue for an additional 6 cycles. PROSTVAC-F will be given as a subq injection on Day 1 of each cycle. Atezolizumab will be given as an infusion on Day 1 of each cycle.
  Other Names: PROSTVAC; Atezolizumab

SUMMARY:
This study is a prospective, open label, single arm phase II trial. A total of 22 patients will be treated with atezolizumab, PROSTVAC, and pre-operative MVA-BN-Brachyury to confirm the efficacy of prostatic combination immunotherapy and to measure the relative change in the number of tumor infiltrating CD8+ lymphocytes within the prostate tissue between the paired biopsy and radical prostatectomy specimens.

DETAILED DESCRIPTION:
Here we propose to use a combination of both checkpoint therapy with dual vaccine therapy. Patients will be treated with an intraprostatic injection of MVA-BN-Brachyury and subcutaneous PROSTVAC therapy. MVA-BN-Brachyury is a replication-deficient, attenuated vaccinia virus (Ankara strain) expressing both a CD8+ T-cell epitope from the brachyury protein and a triad of T-cell co-stimulatory molecules (B7.1, ICAM-1 and LFA-3). MVA-brachury-TRICOM, upon infection of cells, causes innate and then adaptive immune responses, antigen cascade, and improved T cell trafficking to the tumor. Vaccine therapy is one strategy that might increase immune infiltration into the tumor microenvironment. Prostate cancer is known to have minimal lymphocyte infiltration within the microenvironment.

This vaccine strategy of direct injection into the tumor in combination with checkpoint inhibitors has previously been performed in early phase clinical trials.6 Furthermore, this approach of potent vaccine vector use can induce systemic effects as seen in a recent clinical trial of 12 patients with metastatic melanoma.12 In that study, responses were also observed in non-target lesions. In this case, MVA-BN-Brachyury is preferred as in intralesional injection agent over other vaccines due to the increased immunogenicity of MVA compared with fowlpox and improved safety profile for direct injection when compared with vaccinia, due to replication incompetence. In the prior study with MVA-BN-Brachyury no patients were observed to have replication of the virus.

T cell mediated tumor cell killing is dependent on specific T cell recognition of a tumor target antigen, localization of those specific T cells to the tumor, and those T cells properly functioning within the tumor microenvironment. We hypothesize that these three primary issues comprise the major causes of most patients receiving no benefit from checkpoint inhibitor therapy or with vaccine monotherapy. We hypothesize that these issues can be addressed with an active intratumoral virus administration approach combined with the use of a subcutaneously administered vaccine (PROSTVAC) to induce PSA-specific T cell activation in combination with a checkpoint inhibitor. Combination viral based vaccine plus immune checkpoint inhibitor therapy will result in exposure of cancer specific antigens and induce inflammation at the site of the cancer ultimately resulting in significant clinical antitumor effect. Additionally, we hypothesize that the concurrent administration of anti-PD-1 moncolonal antibody therapy is necessary to allow those active T cells to achieve tumor cell killing, and significant overall clinical efficacy.

The addition of atezolizumab is likely to provide additional efficacy over vaccine therapy alone. This is suggested by the induction of PD-1+ T-cells with vaccines.17 Additionally, PD-1 inhibition with nivolumab18 and pembrolizumab19 have shown clinical activity in metastatic prostate cancer. We suggest that the combination will provide even greater efficacy.

Multiple studies have demonstrated a strong correlation between density of lymphocytes and prognosis, including overall survival.13-16 Given the very low density of infiltrating lymphocytes historically in prostate cancer, (Kaur HB, Hum Path 2019) we suggest that the primary endpoint of the change in CD8+ density is a reasonable pharmacodynamic endpoint for this exploratory, hypothesis generating study. However, as this study will be the first to date of the treatment combination, safety will also serve as a co-primary endpoint. The secondary objectives of PSA responses will help confirm the clinical utility of this approach in this target population.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥ 18 years.
* Clinical staged unfavorable intermediate, high-risk or very high-risk prostate cancer per NCCN guidelines.
* Histologically proven prostate adenocarcinoma
* Patient must be a surgical candidate
* ECOG Performance Status ≤ 1.
* Adequate organ function as defined as:

  * Hematologic:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (without granulocyte colony-stimulation factor support within 2 weeks of screening blood test)
* Platelet count ≥ 100 × 109/L (without platelet transfusion within 2 weeks of screening)
* Hemoglobin ≥ 9 g/dL (may not have been transfused within 2 weeks of study treatment initiation)
* White blood cell count (WBC) ≥ 2.5 × 109/L.

  * Hepatic:
* Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) (≤ 3 × ULN for subjects with Gilbert's disease)
* AST and ALT levels ≤ 2.5 × ULN. Patient with a history of unconjugated hyperbilirubinemia with otherwise acceptable liver enzyme levels (as per above criteria) may have higher bilirubin levels.

  * Renal:
* Urine protein/creatinine ratio (UPCR) ≤ 2 mg/mg (≤ 113.2 mg/mmol) UPCR can be calculated with either a random spot urine test or a 24 hour test. The 24-hour urine collection test is more accurate, so it is the definitive test if there is a discrepancy between the urnialysis and the UPCR. A 24-hour urine test is not required, but may be obtained.
* Serum creatinine ≤ 2.0 × ULN or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault equation.
* Highly effective contraception for male subjects throughout the study and for at least 6 months after last study treatment administration if the risk of conception exists.
* Patients must have archival prostate biopsy tissue available with identified prostate cancer. If none is available, a repeat prostate biopsy is mandatory to be eligible for this study. The repeat biopsy if performed must have documented prostate adenocarcinoma. The archival tissue must not have been obtained more than 4 months before enrollment.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Prostate MRI must be performed within the past 8 months.

Exclusion Criteria:

* Prostate cancer histology other than adenocarcinoma.
* Previous treatment for prostate cancer.
* Metastatic disease on imaging (CT, MRI, or NM bone scan) or through tissue biopsy. This includes nodal metastatic disease. A biopsy is not required to rule out metastasis.
* Use of immunosuppressive medication within 28 days of study treatment initiation, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
* Known history of and/or active autoimmune disease requiring systemic treatment. Patients with diabetes mellitus, thyroid disease, vitiligo, or other diseases determined to be not clinically meaningful (per the treating physician) will not be excluded for these conditions.
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent per treating physician's clinical judgment. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid diseases, or other conditions are eligible as per 5.2.5.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  o Cardiovascular disorders:
* Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias within 3 months of study enrollment.
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 180 mm Hg systolic or > 120 mm Hg diastolic despite optimal antihypertensive treatment within 2 weeks of starting treatment.
* Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before first dose.

  * Uncontrolled tumor-related pain.
  * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
  * Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium >ULN).
  * Active Tuberculosis
* Prior allogeneic stem cell or solid organ transplantation.
* Known history of acquired immunodeficiency syndrome.
* Prior or concurrent malignancy whose natural history or treatment, in the opinion of the enrolling investigator, may have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening. Patients with a history of HBV or HCV infection are eligible if the viral load is documented as undetectable at screening. Screening tests for HBV, HCV or HIV are not mandatory by the study but will be performed per the discretion of the study investigators.
* Known history of atopic dermatitis or active skin condition (acute chronic, or exfoliative) that disrupts the epidermis that is clinically significant less than or equal to 180 days before study enrollment.
* Known history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Known history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Live, attenuated (e.g., FluMist) and inactive vaccinations within 28 days of study treatment initiation. Live, attenuated vaccinations are generally discouraged for the duration of the investigational treatment phase of the study. Inactive vaccinations are acceptable after the prostatectomy is performed but cannot be given within 1 week of the study vaccine administration. Live vaccinations require PI approval.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v 5.0 Grade ≥ 3).
* Known allergy to eggs, egg products, or aminoglycoside antibiotics (for example gentamicin or tobramycin).
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
* Known allergy or hypersensitivity to any component of the PROSTVAC or MVA-BN-Brachyury formulation.
* Subjects taking prohibited medications as described in Section 6.6. A washout period of prohibited medications for a period of at least 14 days or as clinically indicated should occur prior to the start of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
To measure the relative change in the number of infiltrating CD8+ lymphocytes within the prostate tissue between the paired biopsy and radical prostatectomy specimens. | Within 8 weeks after cycle2 day 1 visit
  CD8+ lymphocytes in diagnostic biopsy and prostatectomy tissue samples will be quantified by immunohistochemistry (IHC) and analyzed using digital quantification. The relative change will be reported.
To assess the safety of combination immunotherapy in localized prostate cancer through evaluation of Adverse Events (AEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) | Lead-in safety evaluation for first 6 subjects is the time from Cycle 1 Day 1 until the start Cycle 3 Day 1(about 63 days) then continuing through completion of the study. From enrollment through completion of the study for the remaining participants
  Adverse Events (AEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) as characterized by type, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0), timing, seriousness, and relationship to study treatment will be documented.

SECONDARY OUTCOMES:
To assess the undetectable PSA rate | 6 and 12 months
  Undetectable PSA rates at 6 months and 12 months post-prostatectomy. This will be compared with Huntsman Cancer Institute (HCI) historical controls. Matching will be based on NCCN risk categories, age and follow up time.
Assess clinical activity of perioperative combination immunotherapy. | PSA evaluation will occur every 3 months after completion of the adjuvant treatment period. PSA relapse-free survival will be calculated and compared to HCI matched historical controls. Patients will be followed for 2 years after prostatectomy.
  PSA evaluation will occur every 90 days after completion of the adjuvant treatment period. PSA relapse-free survival will be calculated and compared to HCI matched historical controls. Patients will be followed for 2 years after prostatectomy. PSA progression will be defined based on Prostate Cancer Working Group 3 (PCWG3) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No